CLINICAL TRIAL: NCT04938479
Title: D-dimer Prognostic Marker of Cerebral Infarction After Revascularization Procedure
Acronym: D-Dimer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0159
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cerebral Infarction; Cerebral Infarction Recovery
Keywords: Cerebral Infarction; cerebral infarction recovery
MeSH Terms: conditions — Cerebral Infarction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — D-Dimer measurement in blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood sample — D-dimer measurement in blood sample

SUMMARY:
Cerebral infarction is the leading cause of acquired disability in adults. Absence of biological marker used in current practice and identified as a prognostic factor for recovery. D-dimers are degradation products of stabilized fibrin translating an activation of coagulation whatever the cause. Studies have shown that increased D-dimer levels in patients with MI is associated with a higher mortality rate, the link with post-intervention non-revascularization has been demonstrate.

The purpose of this project is to search for a correlation between the level of D-dimer and the degree of recovery evaluated by the NIHSS score

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65
* Cerebral infarctions undergoing a revascularization procedure by thrombolysis and / or thrombectomy, at the Amiens University Hospital between January 2015 and December 2020.
* Patients having benefited from a D-dimer assay (during their stay)

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients under 65 years of age who have presented a heart attack brain and undergoing a revascularization procedure
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between D-dimer concentration and NIHSS score | 3 months
  NIHSS score is based on the clinical neurological examination of the patient. Validated by the scientific community of vascular neurology, among other things in projective clinical research. This score has high inter-observer reproducibility Expressed quantitatively on a scale of 0 to 42 for the NIHSS score A high value of the NIHSS score indicates poor recovery.
Correlation between D-dimer concentration and NIHSS score | 6 months
  NIHSS score is based on the clinical neurological examination of the patient. Validated by the scientific community of vascular neurology, among other things in projective clinical research. This score has high inter-observer reproducibility Expressed quantitatively on a scale of 0 to 42 for the NIHSS score A high value of the NIHSS score indicates poor recovery.
Correlation between D-dimer concentration and the Rankin score | 3 months
  Rankin Scale collected by the neurologist in consultation 3-6 months post stroke.
  Expressed quantitatively on a scale of 0 to 6 for the Rankin scale. A high value of the Rankin scale indicates poor recovery.
Correlation between D-dimer concentration and the Rankin score | 6 months
  Rankin Scale collected by the neurologist in consultation 3-6 months post stroke.
  Expressed quantitatively on a scale of 0 to 6 for the Rankin scale. A high value of the Rankin scale indicates poor recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No